CLINICAL TRIAL: NCT02246816
Title: A Phase 3, Open Label Extension Study for Subjects That Complete Study MP-101-CL-001
Brief Title: A Open Label Extension Study for Subjects That Complete Study MP-101-CL-001
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Transfer of IND to different marketing authorization representative.
Sponsor: Marathon Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-101-CL-002OLE
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-11

CONDITIONS: Short Bowel Syndrome; Short Gut Syndrome; SBS; Short Gut
Keywords: Short Bowel Syndrome; SBS; Chronic Diarrhea; Short Bowel; Short Gut; Short Gut Syndrome; Anti-Diarrheal; Opium Tincture; loperamide; diphenoxylate; ileostomies; tincture of opium; DTO; codeine; morphine; opiate
MeSH Terms: conditions — Short Bowel Syndrome

ARMS (1):
- All Subjects (Experimental): Assigned to receive open-label 0.6 mL, MP-101 (10 mg/mL, Opium Tincture (OT)), USP (Deodorized)
  Interventions: Drug: 0.6 mL, MP-101 (10 mg/mL, Opium Tincture (OT)), USP (Deodorized)

INTERVENTIONS:
Drug: 0.6 mL, MP-101 (10 mg/mL, Opium Tincture (OT)), USP (Deodorized) — 0.6 mL, MP-101 (10 mg/mL, Opium Tincture (OT)), USP (Deodorized)

SUMMARY:
MP-101 will be evaluated in this study to see if it is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female adults, 18 years of age or older
* Have SBS that is inadequately controlled on current antidiarrheal medication (e.g., loperamide or diphenoxylate), including subjects with ileostomies
* Must have been deemed a completer of study protocol MP-101-CL-001.
* Males or non-pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study. Postmenopausal is defined as at least 12 months of natural spontaneous amenorrhea, or at least 6 weeks following surgical menopause (bilateral oophorectomy)
* Females of childbearing potential must agree to use 1 of the following acceptable birth control methods:

  * Surgically sterile (hysterectomy or bilateral oophorectomy)
  * Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation)
  * Intrauterine device (IUD) in place for at least 3 months
  * Abstinence (not having sexual intercourse)
  * Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening and through study completion
  * Stable hormonal contraceptive for at least 3 months prior to study and through study completion
  * Vasectomized partner
* Females of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at Visit 1.
* Be able to understand and provide signed informed consent

Exclusion Criteria:

* Have any history of or active neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, or metabolic disease that is considered clinically significant, is not currently controlled by medication, and is stable as deemed by the Investigator
* Are currently taking antibiotics for bacterial overgrowth
* Have known or suspected pregnancy, planned pregnancy, or lactation
* Have a planned surgery during the course of the study
* Have a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 120 Days

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Cleveland Clinic, Cleveland, Ohio
  - Regional Infectious Disease Infusion Center, Lima, Ohio
  - Vanderbilt Center for Human Nutrition, Nashville, Tennessee